CLINICAL TRIAL: NCT01117246
Title: Pilot Study for the Treatment of Bone Metastases by High Intensity Focused Ultrasound Guided by MRI to Perform Pain Palliation
Brief Title: Pilot Study for Palliation of Pain in Bone Metastases by MR-HIFU
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 998771A; 2010-A00353-36 (Other: CPP sud-ouest et outre mer III)
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Secondary Malignant Neoplasm of Bone
Keywords: bone metastasis; pain palliation
MeSH Terms: interventions — High-Intensity Focused Ultrasound Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated bone metastasis (Experimental): Patients with bone metastasis causing pain.
  Interventions: Device: High Intensity Focused Ultrasound

INTERVENTIONS:
Device: High Intensity Focused Ultrasound — HIFU is the use of focused ultrasound energy to penetrate through soft tissue and causes localized high temperatures (55°C to 70°C) for a few seconds within the target producing well defined regions of protein and nerve denaturation, irreversible cell damage, and coagulative necrosis.
  Other Names: • HIFU; • Ablation; • High Intensity Focused Ultrasound

SUMMARY:
This study is to confirm the safety and technical of MRI guided High Intensity Focused Ultrasound (HIFU) for Palliation for Pain of Skeletal Metastases.

MRI guided high intensity focused ultrasound uses ultrasound to heat and thermally ablate tissue. The MRI system identifies the ultrasound path and monitors heat rise in the tissue. The goal of the study is to show treatment safety and effectiveness. MR-guided HIFU will be performed in patients who pass inclusion/exclusion criteria.

DETAILED DESCRIPTION:
Bone is the third most common site of metastases spread after the liver and the lungs, with a great incidence in breast, prostate, lung, kidney and thyroid cancers. For example, 90% of patients dying from breast cancer and most of patients with advanced prostate cancer suffer from bone metastases, which are frequently responsible of chronic pain and lead to an increase in morbidity and mortality with pathological fractures, compression syndrome and hypercalcemia..Moreover, the increasing longevity of patients with cancer resulting from the improvement of the effectiveness of the treatments leads to a higher incidence and prevalence of metastating bone lesions.

Palliative treatment with management of pain and improvement of quality of life remains the first goal of therapy. Current treatments options include systemic drug therapy (chemotherapy, hormonal therapy, analgesics and bi-phosphonates), local invasive treatment (surgery), local mini-invasive treatment with interventional radiological techniques (cimentoplasty, cryotherapy and radiofrequency ablation) and radiation therapy.

External-beam radiation therapy remains the current standard of care for patients with bone metastases in first intention. However, up to 20-30 % of patients treated do not experience pain relief and recurrence of pain appear in 27 % after treatment. Moreover radiation treatment is limited due to accumulation of dose. Since few years, cryotherapy and percutaneous radiofrequency ablation have shown good results in management of pain with bone metastases, however these techniques are still invasive.

In MRI-guided High Intensity Focused Ultrasound (HIFU), the ultrasound generated by the transducer is focused into a small focal tissue volume at specific target locations. During treatment, the beam of focused ultrasound energy penetrates through soft tissue and causes localized temperatures elevation up 55-70°C for a few seconds within the target producing well defined regions of irreversible protein denaturation, cell damage, and coagulative necrosis. A single exposure of focused ultrasound energy is called a "sonication." Multiple sonications are necessary to ablate the targeted tissue. Tight focusing is designed to limit the ablation to the targeted location.

Applying HIFU energy to a patient's lesion requires treatment planning, targeting of the ultrasound (US) beam to desired locations and monitoring of the energy delivery. In some applications this can be performed using diagnostic ultrasound imaging in combination with the HIFU. While diagnostic US provides some anatomical details and helps with procedure planning and treatment targeting, it does not provide 3D planning, means of measuring the temperature increase generated by HIFU, or metrics for quantifying the energy/dose delivered to the treatment zone. Currently, only MR imaging can provide a validated non-invasive temperature measurement and thermal dose quantification in the treated tissue. Furthermore, these real-time MR temperature measurements can be used to control the HIFU system to deliver optimal temperatures to the target locations. The Philips MR-guided focused ultrasound system will provide real-time tissue temperature mapping in multiple planes and control of the temperature delivering dose to the target location. Recent advances in MR temperature mapping make it possible to achieve temperature accuracy of 1°C in stationary soft tissues.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged > 18 years
* Covered by social security insurance
* Patient able to give consent and able to attend
* study visit
* Weight < 140kg
* Patient with bone metastases
* Pain localized on bone metastases to be treated with NRS (0-10 scale) pain score 4 irrespective of medication
* Targeted tumor accessible for MR-HIFU treatment
* The maximum size of the bone metastases smaller than 8cm in diameter
* Targeted tumor visible by non contrast MRI
* Interface between bone and skin deeper than 10 mm
* Able to communicate sensation during treatment
* Treatment day must be planned at least 2 weeks after any treatment of the primary tumor, chemotherapy or RT treatment of a bone targeted for HIFU

Exclusion Criteria:

* Person subject to a judicial safeguard order, subject participating in another research study including an exclusion period which has not expired at the time of screening
* Patient enrolled in another clinical study related to bone metastases or pain relief treatment
* Pregnant or nursing woman
* Need of surgical stabilization or site at risk of
* fracture
* More than one painful lesion per treatment
* Patients who are not able to tolerate required stationary position during treatment
* HIFU targeted tumor in contact with hollow viscera
* Targeted tumor less than 1 cm to nerve bundles, bladder and bowel
* Targeted tumor located in skull, spine (excepted sacrum) or sternum.
* MRI or contrast agent contraindicated
* Severe Cardiovascular, neurological, renal or hematological chronic disease
* Active infection
* Scar in the beam path
* Orthopedic implant at the site of treatment
* Previous surgery at the site of treatment Patient history, MRI exam
* Primary musculoskeletal malignancies, lymphoma, or leukemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Technical efficacy by medication and pain score | 0, 2, 7, 14, 30, 90 days
  Technical efficacy of HIFU for treatment of bone metastasis as assessed by a change in the medication and pain scores
Safety of treatment | 0-90 days
  Safety of HIFU for treatment of the bone metastasis as determined by adverse event reporting
Safety determined by intended lesions | 0-90 days
  Safety of HIFU for treatment of the bone metastasis as determined by formation of intended lesions.

SECONDARY OUTCOMES:
Treatment size | 0-90 days
  MR-HIFU treatment size measurements
X-Ray treatment size measurements | 0-90 days
  X-Ray treatment size measurements
Length of Hospital Stay | 0-90 days
  Length of Hospital Stay
Quality of Life | 0, 7, 14, 30, 90 days
  Quality of Life Questionnaire scores

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Trillaud, Professor, Principal Investigator — Hôpital St. André, Service de Radiologie
Locations (1):
- Hôpital St. André, Bordeaux, France

REFERENCES:
- [Background] Chow E, Wu JS, Hoskin P, Coia LR, Bentzen SM, Blitzer PH. International consensus on palliative radiotherapy endpoints for future clinical trials in bone metastases. Radiother Oncol. 2002 Sep;64(3):275-80. doi: 10.1016/s0167-8140(02)00170-6. PMID 12242115